CLINICAL TRIAL: NCT00001549
Title: Diagnosis and Natural History Protocol for Patients With Neurological Conditions
Brief Title: Diagnosis and Natural History Study of Patients With Neurological Conditions
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960009; 96-N-0009
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Alzheimer's Disease; Dementia; Movement Disorder; Multiple System Atrophy; Parkinson's Disease
Keywords: Movement Disorders; Parkinson's; Alzheimer's; Screening; Diagnostic Puzzles; Alzheimer Disease; Progressive Supranuclear Palsy; PSP; Restless Leg Syndrome; RLS; Parkinsonism; PD
MeSH Terms: conditions — Alzheimer Disease; Dementia; Movement Disorders; Multiple System Atrophy; Parkinson Disease; Supranuclear Palsy, Progressive; Restless Legs Syndrome; Parkinsonian Disorders

SUMMARY:
The purpose of this study is to improve understanding of neurological conditions. Patients participating in this study will continue receiving medical care, routine laboratory tests, and diagnostics tests (X-rays, CT-scans, and nuclear imaging), from their primary care physician. Doctors at the NIH plan to follow these patients and offer advice and assistance to their primary care physicians.

DETAILED DESCRIPTION:
The objective of this protocol is to provide diagnosis and follow Experimental Therapeutics Branch (ETB) patients not currently entered on another research protocol. No investigational treatments will be administered on this protocol, and the NIH physicians will be playing largely a consultative role to the patient's primary physician.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients may be included on this protocol if they have an identifiable neurological disorder or represent a diagnostic puzzle. These disorders would include patients with Parkinson's disease, Alzheimer's disease, multiple system atrophy, progressive supranuclear palsy, restless legs syndrome, other cognitive and movement disorders, and diagnostic puzzles.

Patients 18-90 years of age, inclusive, are eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 1995-10; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States